CLINICAL TRIAL: NCT00802074
Title: A Randomized, Open-Label, Six-Period, Drug Interaction Study to Assess Steady-State Plasma Amprenavir (APV) and Raltegravir (RTG) Pharmacokinetics Following Administration of RTG 400 mg BID for 14 Days Alone and in Combination With 14 Days of Either Fosamprenavir (FPV) 1400 mg BID, FPV 700 mg BID + RTV 100 mg BID or FPV 1400 mg + RTV 100 mg QD in Healthy Adult Subjects When Under Fasting Conditions
Brief Title: An Interaction Study to Assess Drug Levels in Fasting Healthy Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garden State Infectious Disease Associates, PA (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: COL112775
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Healthy Subjects; Pharmacokinetics study; Pharmacokinetics of medications
MeSH Terms: interventions — Raltegravir Potassium; fosamprenavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A (Active Comparator): Period 1-Raltegravir 400mg BID Period 2- Fosamprenavir 1400mg BID Period 3- Fosamprenavir 1400mg BID + Raltegravir 400mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir
- Group B (Active Comparator): Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg BID + Raltegravir 400mg BID Period 3 Fosamprenavir 1400mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir
- Group C (Active Comparator): Period 1-Raltegravir 400mg BID Period2- Fosamprenavir 700mg BID + Ritonavir 100mg BID Period 3- Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir; Drug: Ritonavir
- Group D (Active Comparator): Period 1-Raltegravir 400mg BID Period 2- Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 700mg BID + Ritonavir 100mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir; Drug: Ritonavir
- Group E (Active Comparator): Period 1-Raltegravir 400mg BID Period 2- Fosamprenavir 1400mg QD + Ritonavir 100mg QD Period 3- Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir; Drug: Ritonavir
- Group F (Active Comparator): Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID Period 3-Fosamprenavir 1400mg QD + Ritonavir 100mg QD
  Interventions: Drug: Raltegravir; Drug: Fosamprenavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Raltegravir — 400mg BID
  Other Names: Isentress; MK-0518
Drug: Fosamprenavir — 1400mg BID, 700 mg BID or 1400 mg QD
  Other Names: Lexiva
Drug: Ritonavir — 100 mg BID or QD
  Other Names: Norvir
  Arms: Group C; Group D; Group E; Group F

SUMMARY:
To date, no study has investigated whether there is a drug interaction between the protease inhibitor fosamprenavir and the integrase inhibitor raltegravir. COL112775 is a randomized, open-label, 6-arm, 3-period, drug interaction study to assess steady-state plasma amprenavir (APV) and raltegravir (RTG) pharmacokinetics in 48 healthy, fasting, HIV-negative adults after administration of a 7-day regimen of RTG 400mg BID alone and after 14-day regimens of unboosted fosamprenavir (FPV) 1400mg twice daily (BID), FPV 700mg/RTV 100mg BID, or FPV 1400mg/ritonavir (RTV) 100mg once daily (QD) with and without concurrent RTG 400mg BID. Blood samples for drug concentration measurement will be collected over 12 hours at the end of each dosing period. Subjects will undergo a physical examination, complete blood count (CBC) with differential, HIV test, hepatitis B/C test, liver function test, renal function analysis, and lipid panel at screening, and all of these tests, except those for HIV and hepatitis B/C, will be repeated at follow-up post-study. Adverse events and adherence (by pill count and medication diary) will be assessed by the investigator/study personnel at the end of each dosing period

DETAILED DESCRIPTION:
This randomized, open-label, six-arm, three-period drug interaction study will recruit 48 healthy volunteers so as to obtain a minimum of 36 evaluable subjects at a single study center in the U.S. The study will have a screening visit, 3 treatment visits for pharmacokinetics (PK) sampling and a follow-up visit. The screening visit will be conducted within 30 days prior to receiving the first dose. Subjects will then be randomized into 1 of 6 treatment groups as shown below:

Cohort Size Period 1 Period 2 Period 3 Sample Days 1 to 7 Days 1-14 Days 1-14

A 8 RTG 400mg BID, FPV 1400mg BID, FPV 1400mg BID + RTG 400mg BID

B 8 RTG 400mg BID, FPV 1400mg BID + RTG 400mg BID , FPV 1400mg BID

C 8 RTG 400mg BID, FPV 700mg BID + RTV 100mg BID, FPV 700mg BID + RTV 100mg BID + RTG 400mg BID

D 8 RTG 400mg BID, FPV 700mg BID + RTV 100mg BID + RTG 400mg BID, FPV 700mg BID + RTV 100mg BID

E 8 RTG 400mg BID, FPV 1400mg QD + RTV 100mg QD, FPV 1400mg QD + RTV 100mg QD + RTG 400mg BID

F 8 RTG 400mg BID, FPV 1400mg QD + RTV 100mg QD + RTG 400mg BID, FPV 1400mg QD + RTV 100mg QD

Study subjects will enter the clinic in the morning prior to dosing in a fasting state and remain at the center for 12 hours following each dose. Fourteen to 21 days following completion of the third dosing period, study subjects will return to the clinic for follow-up assessment. The total duration of the study will be approximately 86 days from screening through follow up. Blood samples for drug concentration measurement of amprenavir (APV) and raltegravir (RTG) concentrations will be collected over 12 hours at the end of each dosing period (at 0 [baseline], 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose). Subjects will undergo a physical examination, CBC with differential, HIV test, hepatitis B/C test, liver function test, renal function analysis, and lipid panel at screening, and all of these tests except those for HIV and hepatitis B/C will be repeated at follow-up post-study. Adverse events and adherence (by pill count and medication diary) will be assessed by the investigator/study personnel at the end of each dosing period. Evaluable patients will be required to have adhered to at least 95% of their study drug doses. Plasma APV concentrations will be analyzed using a validated high-performance liquid chromatography method with tandem mass spectrometric detection (HPLC/MS/MS) and plasma RTG concentrations by triple quadruple mass spectrometry. Plasma APV and RTG pharmacokinetic parameters measured will include maximum concentration (Cmax), time to maximum concentration (Tmax), minimum concentration (Cmin), and area under the concentration-time curve (AUC). All these parameters, except Tmax, will be log-transformed before statistical analysis. Analysis of variance, considering treatment as a fixed effect and subject as a random effect will be performed using Statistical Analysis Software (SAS), and assuming a treatment ratio for steady-state APV PK parameters as 1.0, the 90% confidence intervals will be within the range 0.81-1.24

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no clinically significant abnormality identified by physician by evaluation of medical history, physical examination, clinical laboratory tests or vital signs.
* Between 18 and 64 years.
* A female subject is eligible to participate if she is neither pregnant nor lactating, and falls into one of the following categories:

  * non-childbearing potential including females with documented (medical report verification) hysterectomy or bilateral oophorectomy, or post-menopausal females defined as being amenorrheic for greater than 1 year and having estradiol and follicle stimulating hormone (FSH) levels consistent with menopause.
  * childbearing potential with a negative serum pregnancy test at screen and who agrees to use one of the following methods of contraception from screening or at least two weeks prior to the first dose (whichever is earlier) until the follow-up visit (any contraception method must be used consistently and correctly, i.e., in accordance with both the product label and the instructions of a physician).
* Agreement for complete abstinence from intercourse.
* Double barrier contraception (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide).
* Any intrauterine device (IUD) with published data showing that the expected failure rate is less than 1% per year (not all IUDs meet this criterion)
* Any other method with published data showing that the lowest expected failure rate for that method is less than 1% per year.
* Adequate renal function (calculated creatinine clearance via Cockcroft and Gault method (CrCl) > 50 mL/min).
* Adequate hepatic function (total bilirubin < 2.5mg/dL; hepatic transaminases < 5x normal).
* Adequate hematologic function (absolute neutrophil count [ANC] > 750 neutrophils/mm^3; platelets > 50,000/mm^3; hematocrit > 25%).
* Non-smoker, defined as not having used nicotine-containing products within the past 6 months.
* Willingness and ability to adhere to treatment and follow-up procedures.
* The ability to understand and sign a written informed consent form.
* Body weight > or =50 kg for males and > or=45 kg for females and body mass index (BMI) in the range of 19 to 30 kg/m^2 (BMI = weight [kg]/(height [m])^2).

Exclusion Criteria:

* Have an active infection that required parenteral antibiotics or hospitalization within 2 weeks prior to enrollment.
* A history of or documented gastrointestinal diseases that impact drug absorption.
* Have a significant documented sulfa allergy (e.g., Stevens-Johnson Syndrome) or a history of sensitivity to any of the study medications, or components thereof.
* HIV, Hepatitis B or C positive .
* Cigarette/cigar/pipe smokers.
* History of alcohol/drug abuse or dependence within 12 months of the study, or a history of alcohol consumption in the past six months exceeding 7 units/week for women and 14 units/week for men (where 1 unit = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor).
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Use of prescription or non-prescription drugs (including aspirin and nonsteroidal anti-inflammatory drug (NSAIDs), vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer, such as St. John's Wort) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator the medication will not interfere with the study procedures or compromise subject safety.
* Subjects who have donated plasma within 7 days prior to the screening visit or where participation in this study would result in donation of blood in excess of 500 mL of blood within 56 day period.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David V Condoluci, DO, Principal Investigator — GSIDA
Locations (1):
- Garden State Infectious Disease Associates, PA, Voorhees Township, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group E: Period 1-Raltegravir 400mg BID Period 2- Fosamprenavir 1400mg once daily (QD) + Ritonavir 100mg QD Period 3- Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Started | 9 | 8 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 6 | 7 | 7 | 7
Not Completed | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Total
Number analyzed (Participants) | 7 | 7 | 6 | 7 | 7 | 7 | 41
Age, Customized [Number; unit: participants]
  18-25 | 4 | 4 | 3 | 3 | 3 | 3 | 20
  26-33 | 2 | 0 | 2 | 1 | 4 | 3 | 12
  34-41 | 0 | 2 | 1 | 1 | 0 | 0 | 4
  42-49 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  50 and older | 0 | 1 | 0 | 1 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 2 | 3 | 4 | 18
  Male | 4 | 3 | 4 | 5 | 4 | 3 | 23
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 6 | 7 | 7 | 7 | 41

OUTCOME MEASURES:

1. Primary Outcome: Cmin/Cmax: Fasting Steady-state Plasma Amprenavir (APV) Pharmacokinetics (PK) Following Admin of Fosamprenavir (FPV) 1400mg BID, FPV 700mg/Ritonavir (RTV) 100 mg BID, or FPV 1400mg/RTV 100mg QD With and Without Concurrent Raltegravir (RTG) 400mg BID.
Description: Amprenavir (APV) is the active ingredient/metabolite of Fosamprenavir (FPV). APV minimum concentration (Cmin), maximum concentration (Cmax), area under the plasma concentration-time curve (AUC), and oral clearance (CL/F) as determined from APV concentrations observed in blood samples obtained at baseline, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours during the BID regimens (FPV 1400mg BID, FPV 700mg/RTV 100 mg BID), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours during the QD regimen (FPV 1400mg/RTV 100mg QD). As Groups A and B received the same regimens (albeit in different order), PK data for these two groups were collated, then assessed. For the same reason, PK data from Groups C and D regimens were collated before assessment, as were the PK data from Groups E and F.
Time Frame: Day 14 of the FPV 1400mg BID, FPV 1400mg/RAL 400mg BID, FPV 700mg/RTV 100mg BID, FPV 700mg/RTV 100mg/RAL 400mg BID, FPV 1400mg/RTV 100mg QD, and FPV 1400mg/RTV 100mg QD plus RAL 400mg BID regimens
Measure: Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Group A & B: Group A Period 1-Raltegravir 400mg BID Period 2- Fosamprenavir 1400mg BID Period 3- Fosamprenavir 1400mg BID + Raltegravir 400mg BID
  Group B Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg BID + Raltegravir 400mg BID Period 3 Fosamprenavir 1400mg BID
- Group C & D: Group C Period 1-Raltegravir 400mg BID Period2- Fosamprenavir 700mg BID + Ritonavir 100mg BID Period 3- Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID
  Group D Period 1-Raltegravir 400mg BID Period 2- Fosamprenavir 700mg BID + Ritonavir 100mg BID + Raltegravir 400mg BID Period 3-Fosamprenavir 700mg BID + Ritonavir 100mg BID
- Group E & F: Group E Period 1-Raltegravir 400mg BID Period 2- Fosamprenavir 1400mg QD + Ritonavir 100mg QD Period 3- Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID
  Group F Period 1-Raltegravir 400mg BID Period 2-Fosamprenavir 1400mg QD + Ritonavir 100mg QD + Raltegravir 400mg BID Period 3-Fosamprenavir 1400mg QD + Ritonavir 100mg QD
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 14 | 13 | 14
ng/mL
  Cmin (ng/mL) | 0.57 [0.43 to 0.76] | 0.81 [0.58 to 1.13] | 0.50 [0.34 to 0.74]
  Cmax (ng/mL) | 0.73 [0.53 to 1.01] | 0.86 [0.64 to 1.15] | 0.82 [0.67 to 0.99]

2. Primary Outcome: AUC: Fasting Steady-state Plasma Amprenavir (APV) Pharmacokinetics (PK) Following Administration of Fosamprenavir (FPV) 1400mg BID, FPV 700mg/Ritonavir (RTV) 100 mg BID, or FPV 1400mg/RTV 100mg QD With and Without Concurrent Raltegravir (RTG) 400mg BID.
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: ng•h/mL
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 14 | 13 | 14
ng•h/mL | 0.64 [0.47 to 0.88] | 0.84 [0.64 to 1.08] | 0.76 [0.59 to 0.97]

3. Secondary Outcome: Number of Participants Who Experienced Adverse Events
Description: Safety/tolerability data included all adverse events (AEs) reported within the time frame of each regimen evaluated. The intent was to compare AE's for each sequence and not for each regimen. 3The regimens for which AE information was culled were:
  * RAL 400mg BID alone
  * FPV 1400mg BID alone
  * FPV 700mg/RTV 100 mg BID alone
  * FPV 1400mg/RTV 100mg QD alone
  * FPV 1400mg BID combined with RAL 400mg BID
  * FPV 700mg/RTV 100 mg BID combined with RAL 400mg BID
  * FPV 1400mg/RTV 100mg QD combined with RAL 400mg BID The severity of reported AEs was graded according to DAIDS criteria, Version 1.0 (National Institute of Allergy and Infectious Diseases (NIAID). Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0. Division of Acquired Immunodeficiency Syndrome (DAIDS), Washington D.C.; 2004).
Time Frame: Day 0 through Day 49
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Number analyzed (Participants) | 7 | 7 | 6 | 7 | 7 | 7
participants | 3 | 3 | 4 | 4 | 5 | 5

4. Primary Outcome: CL/F: Fasting Steady-state Plasma Amprenavir (APV) Pharmacokinetics (PK) Following Administration of Fosamprenavir (FPV) 1400mg BID, FPV 700mg/Ritonavir (RTV) 100 mg BID, or FPV 1400mg/RTV 100mg QD With and Without Concurrent Raltegravir (RTG) 400mg BID.
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: L/h
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 14 | 13 | 14
L/h | 1.57 [1.14 to 2.16] | 1.05 [0.74 to 1.50] | 1.63 [1.22 to 2.18]

5. Primary Outcome: Cmin/Cmax: Steady-state Plasma RTG PK Following Admin of RTG 400mg BID Alone and Following Co-administration With FPV 1400mg BID, FPV 700mg/RTV 100 mg BID, or FPV 1400mg/RTV 100mg QD
Description: Amprenavir (APV) is the active ingredient/metabolite of Fosamprenavir (FPV). RAL minimum concentration (Cmin), maximum concentration (Cmax), area under the plasma concentration-time curve (AUC), and oral clearance (CL/F) as determined from RAL concentrations observed in blood samples obtained at baseline, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours during the period when RAL 400mg BID was administered with the FPV-Containing BID regimens (FPV 1400mg BID, FPV 700mg/RTV 100 mg BID), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours during the period when RAL 400mg BID was administered with the FPV QD regimen (FPV 1400mg/RTV 100mg QD). As Groups A and B received the same regimens (albeit in different order), PK data for these two groups were collated, then assessed. For the same reason, PK data from Groups C and D regimens were collated before assessment, as were the PK data from Groups E and F.
Time Frame: Day 7 of the RAL 400mg BID regimen and Day 14 of the RAL 400mg/FPV 1400mg BID, RAL 400mg/FPV 700mg/RTV 100mg BID, and RAL 400mg BID Plus FPV 1400mg/RTV 100mg QD regimens
Measure: Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 14 | 13 | 14
ng/mL
  Cmin (ng/mL) | 0.62 [0.43 to 0.89] | 0.64 [0.43 to 0.97] | 0.75 [0.59 to 0.96]
  Cmax (ng/mL) | 0.72 [0.41 to 1.26] | 0.49 [0.25 to 0.97] | 1.06 [0.62 to 1.81]

6. Primary Outcome: AUC: Steady-state Plasma RTG PK Following Administration of RTG 400mg BID Alone and Following Co-administration With FPV 1400mg BID, FPV 700mg/RTV 100 mg BID, or FPV 1400mg/RTV 100mg QD
Description: as for outcome 5
Time Frame: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 14 | 13 | 14
ng*h/mL | 0.63 [0.40 to 0.99] | 0.45 [0.24 to 0.84] | 0.85 [0.54 to 1.33]

7. Primary Outcome: CL/F: Steady-state Plasma RTG PK Following Administration of RTG 400mg BID Alone and Following Co-administration With FPV 1400mg BID, FPV 700mg/RTV 100 mg BID, or FPV 1400mg/RTV 100mg QD
Description: as for outcome 5
Time Frame: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: L/h
Arm/Group | Group A & B | Group C & D | Group E & F
Number analyzed (Participants) | 14 | 13 | 14
L/h | 1.46 [0.92 to 2.2] | 2.00 [1.10 to 3.62] | 1.18 [0.77 to 1.79]

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AE) included events starting on or after Day 0 through Day 49.
Description: If a subject experienced more than 1 of a given AE, the subject is counted only once for that AE.
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 3/7 | 3/7 | 4/6 | 4/7 | 5/7 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=7) | Group B (N=7) | Group C (N=6) | Group D (N=7) | Group E (N=7) | Group F (N=7)
Nausea/Vomiting/Diarrhea (Gastrointestinal disorders) | 1 | 3 | 2 | 4 | 4 | 4
fatigue (General disorders) | 2 | 0 | 0 | 1 | 0 | 1
numbness of lips/tongue/mouth (General disorders) | 1 | 0 | 0 | 1 | 1 | 3
headache/migraine (Nervous system disorders) | 1 | 0 | 0 | 1 | 2 | 1
cold symptoms/uri/fever (General disorders) | 1 | 0 | 1 | 0 | 0 | 1
Itching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
frequent urination (General disorders) | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Data for Primary outcome measure assessments are not available per intervention. Values reported as means are of uncertain measure type (data are no longer available).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No